CLINICAL TRIAL: NCT03439722
Title: Sleep in Cluster Headache: Sleep Parameters in- and Outside a Cluster Bout
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, MD, Ph.d.-student Nunu Lund, MD, Danish Headache Center
Other Study IDs: H-7-2014-020 Sleep study
Record Dates: First submitted 2016-07-27; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Cluster Headache
Keywords: cluster headache; sleep disturbances
MeSH Terms: conditions — Cluster Headache; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Episodic cluster headache patients will be admitted for 1 night where a polysomnography will be performed by the Danish Center of Sleep Medicine.
  Interventions: Other: Polysomnography
- Controls: Controls will be admitted for 1 night where a polysomnography will be performed by the Danish Center of Sleep Medicine.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Participants will be admitted for 1 night at the Danish Center of Sleep Medicine for polysomnography.

SUMMARY:
Sleep study in episodic cluster headache patients.

DETAILED DESCRIPTION:
This is an explorative study that aims to describe the sleep in 30 episodic cluster headache patients in- and outside of cluster using polysomnography. Data will be compared to a group of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years of age
* Episodic cluster headache according to ICHD-III beta
* Ability to differentiate attacks of other primary headaches from cluster headache.
* 1-8 daily attacks
* Cluster bouts normally lasting more than 2 weeks

Exclusion Criteria:

* Treatment with psychiatric medication other than lithium.
* Pregnancy or breastfeeding
* Serious somatic or psychiatric disorders
* Chronic primary or secondary headache
* Alcohol intake higher than 14 units a week for males and 7 units a week for females.
* Cannot accept the conditions of the trial.
* Does not understand Danish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Episodic cluster headache patients diagnosed according to International Classification of Headache disorders III beta (ICHD III beta)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare total sleep time (hours) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients with healthy controls | From study initiation to January 2018
  Compare sleep latency (minutes) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare rapid eye movement sleep latency (hours) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare prevalence of N1 sleep (%) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare prevalence of N2 sleep (%) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare prevalence of N3 sleep (%) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare prevalence of REM sleep (%) during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare arousals/hour of sleep during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare awakenings/hour of sleep during one night of polysomnography using mixed models analyses.
Compare the macrostructure of sleep in episodic cluster headache patients in bout with in remission | From study initiation to January 2018
  Compare apnea-hypopnea index during one night of polysomnography using mixed models analyses.

SECONDARY OUTCOMES:
The presence of any sleep disorders in patients and controls | From study initiation to January 2018
  Cpmpare the same parameters (Primary outcomes 1-11) in patients and controls. Prevalences will be compared using chi-square tests across categories. If n<5 Mann-Whitney U-test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Nunu Lund, MD, Principal Investigator — Danish Headache Center, Rigshospitalet - Glostrup
Locations (1):
- Danish Headache Center, Dept. of Neurology, Rigshospitalet -Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided